CLINICAL TRIAL: NCT05433259
Title: The Influence on Biometric Factors Changes by Different OK Lens
Brief Title: Biometric Factors Changes Caused by Myopia Orthokeratology (OK) Lens
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Yune Zhao, Vice president of Eye Hospital of Wenzhou Medical University, Wenzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: OK lens-Angio OCT
Record Dates: First submitted 2022-06-21; First posted 2022-06-27 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Contact Lenses

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CRT type lens (Experimental): Subjects fitted with CRT type lenses
  Interventions: Device: Overnight orthokeratology
- VST type lens (Experimental): Subjects fitted with VST type lenses
  Interventions: Device: Overnight orthokeratology

INTERVENTIONS:
Device: Overnight orthokeratology — Subjects require to wear the lenses every night, with a recommended time of 6-8 hours.

SUMMARY:
Subjects fit with VST or CRT type lens are reviewed 1 day to 2 year after first wearing the lens. Ocular examinations were performed, including slit-lamp biomicroscope, uncorrected distance visual acuity (UDVA), corrected distance visual acuity (CDVA), corneal topography (Medmont E300W, Medmont Pty Ltd, Melbourne, Australia), corneal refractive power (autorefractometer, KR880, Topcon, JAPAN), corneal epithelial thickness (Optical Coherence Tomography, RTVue-XR), axial length using IOL-Master 700 (Carl Zeiss Meditec AG). To investigate corneal and retina changes caused by overnight OK lens.

ELIGIBILITY:
Inclusion Criteria:

* Normal subjects without any history of ocular surgeries or diseases (except for refractive errors) or systemic diseases that might affect contact lens wearing. The spherical error between -1.0 and -5.0 D, cylindrical error of at most 2.0 D, and a corrected distance visual acuity of 20/20 or better.

Exclusion Criteria:

* Subjects who had previously worn contact lens, were also excluded

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-03-12 (Actual); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
change of Corneal Epithelium | up to 1 day, 1 week,1 month
  All epithelial thickness and treatment zone area record by baseline and follow up examination.

SECONDARY OUTCOMES:
Axial length | up to 2 years
  Axial length growth after lens wear

CONTACTS AND LOCATIONS:
Locations (1):
- Eye Hospital of Wenzhou Medical College, Wenzhou, Zhejiang, China